CLINICAL TRIAL: NCT05300555
Title: Cost-effectiveness Analysis Between Two Anticoagulation Strategies for Atrial Fibrillation in the Postoperative Period of Coronary Artery Bypass Graft Surgery
Acronym: TASK-POAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Jr, PHD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC 5074//20/103
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation New Onset
Keywords: ANTICOAGULANTS; CORONARY ARTERY BYPASS GRAFT; ATRIAL FIBRILLATION; POST OPERATIVE ATRIAL FIBRILLATION; COST-EFECTIVENESS; ANTICOAGULANT THERAPY AFTER NEW ONSET POST OPERATIVE ATRIAL FIBRILLATION
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban group (Experimental): After randomization, the patient will start medication (rivaroxaban 20mg per day or 15mg per day if eGFR between 30 and 50ml/min/1,73m²) within 24 hours. The medication will be prescribed up to 30 days after hospital discharge and if there is no clinical, electrocardiographic and Holter evidence of AF, the medication will be discontinued
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet
- Warfarin group (Experimental): After randomization, the patient will start medication within 24 hours. Bridge with heparin or enoxaparin is recommended. The INR target is between 2,0 and 3,0. The medication will be prescribed up to 30 days after hospital discharge and if there is no clinical, electrocardiographic and Holter evidence of AF, the medication will be discontinued
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban 20 MG Oral Tablet — After randomization, the patient will start medication (rivaroxaban 20mg per day or 15mg per day if eGFR between 30 and 50ml/min/1,73m²) within 24 hours. The medication will be prescribed up to 30 days after hospital discharge and if there is no clinical, electrocardiographic and Holter evidence of AF, the medication will be discontinued
  Other Names: Rivaroxaban
  Arms: Rivaroxaban group
Drug: Warfarin — After randomization, the patient will start medication within 24 hours. Bridge with heparin or enoxaparin is recommended. The INR target is between 2,0 and 3,0. The medication will be prescribed up to 30 days after hospital discharge and if there is no clinical, electrocardiographic and Holter evidence of AF, the medication will be discontinued
  Arms: Warfarin group

SUMMARY:
Coronary artery bypass graft (CABG) surgery is a common intervention in patients with coronary artery disease (CAD). The presence of new postoperative atrial fibrillation / atrial flutter (POAF) occurs in 15-40% of patients undergoing this procedure, with a high rate of complications, including increased hospital length of stay, with a consequent increase in the costs. In addition, the presence of POAF increases the rate of thromboembolic events such as stroke and mortality in the short and long term.

Anticoagulant treatment in patients with atrial fibrillation and atrial flutter (AF) lato sensu is already a well-established therapy in patients at high risk, defined by CHADS-VASC greater than or equal to 2. The use of direct-acting anticoagulants (DOACS) is standard therapy for those patients. In the POAF scenario, there is a recommendation for anticoagulation in high-risk patients for at least 30 days, however, despite being an entity with a poor prognosis in the short and long term, it is an undertreated entity. At present, there is no evidence of anticoagulant treatment of POAF with DOACS, and warfarin is the standard therapy. Warfarin is a drug that needs laboratory control of prothrombin time (PT) and anticoagulation bridge with other anticoagulants, usually using heparin and enoxaparin. We believe that because warfarin is the standard drug in this scenario, it is not prescribed on a regular basis, since it increases costs, length of hospital stay and is less effective than DOACS in AF lato sensu.

Thus, the research project intends to compare the cost-effectiveness, assessed by QALY, related to the warfarin prescription strategy associated with bridge anticoagulation versus the rivaroxaban prescription in patients who presented POAF with a minimum duration of 12 hours or AF that requires intervention. Medications will be started during hospitalization. After randomization, anticoagulant medication will be started within 24 hours. The patient will be reassessed in 30 days and if there is no evidence of maintenance of AF, the anticoagulant medication will be discontinued and the standard treatment for CAD will be maintained. Secondary outcomes will be: clinical outcomes, such as: (1) Death; (2) stroke; (3) myocardial infarction (MI); (4) Readmission; (5) Systemic embolization; (6); Surgical reintervention; (6) Bleeding using the ISTH score; (7) Infection. The safety outcome will be the bleeding assessment according to the bleeding score of the ISTH (International Society on Thrombosis and Haemostasis).

Considering that POAF is a prevalent entity and associated with a worse prognosis in the short and long term, as well as despite recommendations for guidelines to keep these patients anticoagulated, it is noted that the prescription of anticoagulation at hospital discharge is low. Considering that there is no clear evidence in studies on the use of DOAC in this population, we understand that the search for medications that lead to better cost-benefit, as well as better dosage and bleeding rates not lower than the use of warfarin, could lead to a higher rate prescribing anticoagulants for these patients, reducing costs, clinical and mortality outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New atrial/flutter fibrillation / flutter lasting more than 12 hours in the postoperative period of CABG
* Individuals in both sex over the age of 18 years

Exclusion Criteria:

* Inability to sign the free and informed consent form
* Contraindication to anticoagulant therapy
* Renal dysfunction with eGFR less than 30ml / min / 1.73m² or dialysis therapy
* Patients with previous AF
* Pregnancy
* Concomitant valve surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness between rivaroxaban and warfarin group | 30 days after hospital discharge
  The primary outcome will be the cost-effectiveness, assessed by QALY, of the treatments in both therapeutic groups (rivaroxaban and warfarin) during the hospital stay with follow-up for 30 days after hospital discharge.

SECONDARY OUTCOMES:
Bleeding according to ISTH bleeding score | 30 days after hospital discharge
  Security outcome
Secondary outcome | 30 days after hospital discharge
  (1) Death; (2) stroke; (3) MI; (4) Readmission; (5) Systemic embolization; (6); Surgical reintervention; (6) Bleeding using the ISTH score; (7) Infection;

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute - University of São Paulo, São Paulo, São Paulo, Brazil